CLINICAL TRIAL: NCT04092361
Title: Macular and Retinal Changes in Unilateral Amblyopia Using Optical Coherence Tomography
Brief Title: Changes in Amblyopia Using Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alyaa mohamed yousef ahmed elkabsh, principle investigator, Assiut University
Other Study IDs: OCT changes in amblyopia
Record Dates: First submitted 2019-09-07; First posted 2019-09-17 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- anisometropic amblyopia
  Interventions: Device: optical coherence tomography
- strabismic amblyopia
  Interventions: Device: optical coherence tomography
- deprivational amblyopia
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — It generates cross sectional images by analyzing the time delay and magnitude change of low coherence light as it is backscattered by ocular tissues. An infrared scanning beam is split into a sample arm and a reference arm. As the sample beam returns to the instrument it is correlated with the reference arm in order to determine distance and signal change via photodetector measurement. The resulting change in signal amplitude allows tissue differentiation by analysis of the reflective properties, which are matched to a false color scale. As the scanning beam moves across tissue, the sequential longitudinal signals, or A-scans, can be reassembled into a transverse scan yielding cross-sectional images, or B-scans, of the subject. The scans can then be analyzed in a variety of ways providing both empirical measurements (e.g. RNFL or retinal thickness/volume) and qualitative morphological information.

SUMMARY:
There have been multiple trials to investigate the morphological changes in the macula and retinal nerve fiber layer of amblyopic eyes, due to the different published results and the lack of evident association between these changes and the patients' parameters. So, we perform this study to compare the variations in macular parameters (central thickness, average thickness, macular volume) and peripapillary thickness in different cases of amblyopic eyes versus the normal fellow eyes using spectral-domain optical coherence tomography. In addition, to estimate the relationship of optical coherence tomography variations with different defined patients' parameters (age, sex, best corrected visual acuity, spherical equivalent refractive error, and axial length).

DETAILED DESCRIPTION:
Amblyopia remains an important cause of low visual acuity,affecting 2% to 6% of the general population. Unilateral amblyopia is defined as reduced best-corrected visual acuity secondary to an abnormal visual experience during the critical period of visual development. Classic causes include strabismus, anisometropia, form deprivation or a combination of these factors .

The normal postnatal reduction (apoptosis) of retinal ganglion cells is arrested in amblyopia which would cause increase in retinal nerve fiber layer thickness as hypothesized by Yen et al .This also would affect the normal maturation of the macula, including movement of Henle's fibers away from the foveola. This would result in increased foveal thickness. Furthermore, because of the reduced apoptosis of retinal ganglion cells, the thickness of the ganglion cell layer in the macula would also be increased.

Optical coherence tomography : is a non-contact and non-invasive technique that help in assessment of retina abnormalities. The high resolving power (10um - Time Domain, 5um - Spectral Domain) provides excellent detail for evaluating the vitreo-retinal interface, neurosensory retinal morphology, and the retinal pigmented epithelial-choroid complex. It generates cross sectional images by analyzing the time delay and magnitude change of low coherence light as it is backscattered by ocular tissues. An infrared scanning beam is split into a sample arm (directed toward the subject) and a reference arm (directed toward a mirror). As the sample beam returns to the instrument it is correlated with the reference arm in order to determine distance and signal change via photodetector measurement. The resulting change in signal amplitude allows tissue differentiation by analysis of the reflective properties, which are matched to a false color scale. As the scanning beam moves across tissue, the sequential longitudinal signals, or A-scans, can be reassembled into a transverse scan yielding cross-sectional images, or B-scans, of the subject. The scans can then be analyzed in a variety of ways providing both empirical measurements (e.g. retinal thickness/volume) and qualitative morphological information.

ELIGIBILITY:
Inclusion Criteria:

1. Age>16 and <40 years
2. Patients with unilateral amblyopia ( anisometropic , strabismic and deprivational amblyopia ) .

Exclusion Criteria:

1. Age<16 and >40 years.
2. Patients with structural abnormality in their eye , mentally retarded patients .

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all cooperative patients that fulfill inclusion criteria
  1. Age>16 and <40 years
  2. Patients with unilateral amblyopia ( anisometropic , strabismic and deprivational amblyopia )
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
To measure retinal layers and macular thickness changes in cases of unilateral amblyopia using optical coherence tomography in comparison with the other sound eye. | from october 1st 2019 to october 1st 2020
  Foveal thickness (mean thickness in the central 1000-μm diameter area) and central foveal thickness (mean thickness at the point of intersection of 6 radial scans) are 212 ± 20 and 182 ± 23 μm, respectively. Macular thickness measurements were thinnest at the center of the fovea, thickest within 3-mm diameter of the center, and diminished toward the periphery of the macula. The temporal quadrant was thinner than the nasal quadrant.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKee SP, Schor CM, Steinman SB, Wilson N, Koch GG, Davis SM, Hsu-Winges C, Day SH, Chan CL, Movshon JA, et al. The classification of amblyopia on the basis of visual and oculomotor performance. Trans Am Ophthalmol Soc. 1992;90:123-44; discussion 145-8. No abstract available. PMID 1494815
- [Background] Graham PA. Epidemiology of strabismus. Br J Ophthalmol. 1974 Mar;58(3):224-31. doi: 10.1136/bjo.58.3.224. No abstract available. PMID 4834596
- [Background] Kiorpes L, McKee SP. Neural mechanisms underlying amblyopia. Curr Opin Neurobiol. 1999 Aug;9(4):480-6. doi: 10.1016/s0959-4388(99)80072-5. PMID 10448162
- [Background] de Zarate BR, Tejedor J. Current concepts in the management of amblyopia. Clin Ophthalmol. 2007 Dec;1(4):403-14. PMID 19668517
- [Background] Choi MY, Lee KM, Hwang JM, Choi DG, Lee DS, Park KH, Yu YS. Comparison between anisometropic and strabismic amblyopia using functional magnetic resonance imaging. Br J Ophthalmol. 2001 Sep;85(9):1052-6. doi: 10.1136/bjo.85.9.1052. PMID 11520755
- [Background] Yen MY, Cheng CY, Wang AG. Retinal nerve fiber layer thickness in unilateral amblyopia. Invest Ophthalmol Vis Sci. 2004 Jul;45(7):2224-30. doi: 10.1167/iovs.03-0297. PMID 15223799
- [Background] Hee MR, Izatt JA, Swanson EA, Huang D, Schuman JS, Lin CP, Puliafito CA, Fujimoto JG. Optical coherence tomography of the human retina. Arch Ophthalmol. 1995 Mar;113(3):325-32. doi: 10.1001/archopht.1995.01100030081025. PMID 7887846
- [Background] Yoon SW, Park WH, Baek SH, Kong SM. Thicknesses of macular retinal layer and peripapillary retinal nerve fiber layer in patients with hyperopic anisometropic amblyopia. Korean J Ophthalmol. 2005 Mar;19(1):62-7. doi: 10.3341/kjo.2005.19.1.62. PMID 15929489
- [Background] Yakar K, Kan E, Alan A, Alp MH, Ceylan T. Retinal Nerve Fibre Layer and Macular Thicknesses in Adults with Hyperopic Anisometropic Amblyopia. J Ophthalmol. 2015;2015:946467. doi: 10.1155/2015/946467. Epub 2015 May 7. PMID 26064676